CLINICAL TRIAL: NCT06312501
Title: Evaluating the Effectiveness of Remote Patient Monitoring (Satelia® Cardio) for Patients With Heart Failure (TELESAT-HF Study)
Brief Title: Remote Patient Monitoring for Patients With Heart Failure in France
Acronym: TELESAT-HF
Status: Completed | Type: Observational
Sponsor: Satelia (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-0020 TELESAT-HF
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Patient Empowerment; Cardiac Failure
Keywords: Remote patient monitoring; Heart failure; Cardiac decompensation; Telehealth
MeSH Terms: conditions — Heart Failure; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RPM heart failure patients: Patients that use RPM for the follow-ups of their condition.
  Interventions: Device: Satelia®Cardio
- Real-life heart failure patients recieving conventional care: Patients that do not use any medical devices and/or solutions such as RPM for the follow-ups of their condition.
  Interventions: Other: Conventional care

INTERVENTIONS:
Device: Satelia®Cardio — Use of a remote patient monitoring system by NP Medical.
  Groups: RPM heart failure patients
Other: Conventional care — No use of RPM solutions for follow-up
  Groups: Real-life heart failure patients recieving conventional care

SUMMARY:
The goal of this multicenter observational longitudinal cohort study is to evaluate the ability of a Remote Patient Monitoring (RPM) program to prevent cardiac decompensation by detecting weak signals of decompensation early in patients with chronic heart failure in France.

The main question it aims to answer is whether an RPM solution can provide the improvement in overall patient survival

Participants will answer to questionnaires provided by the RPM solution for the follow-up of their condition.

Researchers will compare the following cohorts to see if RPM can improve their condition:

* Cohort 1: using RPM for follow-ups.
* Cohort 2: conventional care and not using any devices and solutions for the follow-ups.

DETAILED DESCRIPTION:
TELESAT study is a national-scale observational prospective cohort study conducted in France from August 2018 to December 2022.

The study was conducted using the French national health data system known as the Système National des Données de Santé (SNDS) which covers approximately 99% of the French population.

ELIGIBILITY:
Inclusion Criteria:

* residing in France
* having heart failure
* adults over the age of 18 years
* New York Heart Association (NYHA) score≥2 and Brain Natriuretic Peptid (BNP)>100 pg/ml or N-terminal pro BNP>1000 pg/ml OR prior hospitalization for heart failure

Exclusion Criteria:

* physician's assessment deemed patient not be physically or mentally able to be remotely monitored
* had chronic dialysis
* severe liver failure
* the presence of any other medical condition resulting in a less than one-year life expectancy,
* an estimated low adherence to treatment
* lack of a stable place of residence
* refusing to participate in the program ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20,000 patients with heart failure across France.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of All Causes Deaths | August 2018 to December 2021
  Number of deaths for any cause

SECONDARY OUTCOMES:
Number of unplanned heart failure Hospitalization | August 2018 to December 2021
  Number of unplanned hospitalization for heart failure
Number of All Causes Deaths in elderly patients | August 2018 to December 2021
  Number of deaths for any cause in the elderly population
Number of unplanned hospitalization for heart failure in elderly patients | August 2018 to December 2021
  Number of unplanned hospitalization for heart failure in elderly patients

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Pages, MD, Study Director — NP Medical
Locations (1):
- NP Medical, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pages N, Picard F, Barritault F, Amara W, Lafitte S, Maribas P, Abassade P, Labarre JP, Boulestreau R, Chaouky H, Abdennadher M, Lemieux H, Lasserre R, Bedel C, Betito L, Nisse-Durgeat S, Diebold B. Remote patient monitoring for chronic heart failure in France: When an innovative funding program (ETAPES) meets an innovative solution (Satelia(R) Cardio). Digit Health. 2022 Aug 22;8:20552076221116774. doi: 10.1177/20552076221116774. eCollection 2022 Jan-Dec. PMID 36034602
- [Background] Jourdain P, Pages N, Amara W, Maribas P, Lafitte S, Lemieux H, Barritault F, Seronde MF, Labarre JP, Chaouky H, Bedel C, Betito L, Nisse-Durgeat S, Picard F. Perceptions and satisfaction of patients with chronic heart failure when using a remote monitoring web application named Satelia(R) Cardio. Ann Cardiol Angeiol (Paris). 2023 Jun;72(3):101606. doi: 10.1016/j.ancard.2023.101606. Epub 2023 May 25. French. PMID 37244215
- [Background] Creton S, Saadi M, Monfort H, Yaghobian S, Pages N, Nisse-Durgeat S, Diebold B. The Clinical Impact and Good Practices of Remote Patient Monitoring for Chronic Heart Failure: A French Case Report. Patient Prefer Adherence. 2024 Jan 16;18:131-135. doi: 10.2147/PPA.S445638. eCollection 2024. PMID 38249685
- See also: Satelia website — http://satelia.eu
- See also: TELESAT study from the data hub — https://www.health-data-hub.fr/projets/tele-sat-evaluation-de-limpact-de-la-telesurveillance-par-le-dispositif-sateliar-cardio